CLINICAL TRIAL: NCT07073794
Title: A Phase 2 Pragmatic Clinical Trial to Evaluate Administration of Cancer Therapy in the Patients' Homes Versus in Clinic in Black Men With Advanced or Metastatic Prostate Cancer
Brief Title: Evaluating In Home Cancer Therapy Versus In Clinic Cancer Therapy in Black Men With Locally Advanced, Biochemically Recurrent and Metastatic Prostate Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC240507; NCI-2025-04662 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-010825 (Other: Mayo Clinic Institutional Review Board); MC240507 (Other: Mayo Clinic); W81XWH-24-1-1106 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Locally Advanced Prostate Carcinoma; Metastatic Prostate Carcinoma; Stage III Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Antineoplastic Protocols; Delivery of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (in clinic treatment, in home treatment) (Experimental): Patients receive standard of care treatment in the clinic for 6-12 weeks then receive treatment in the home with CCBW for 12-24 weeks in the absence of disease progression or unacceptable toxicity. Patients receive any remaining treatment in the clinic.
  Interventions: Drug: Cancer Therapeutic Procedure; Other: Health Care Delivery; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Cancer Therapeutic Procedure — Given standard of care cancer treatment in clinic
  Other Names: anticancer therapy; Cancer Therapy; Cancer Treatment; Malignant Neoplasm Therapy; Malignant Neoplasm Treatment
Drug: Cancer Therapeutic Procedure — Given standard of care cancer treatment in home
  Other Names: anticancer therapy; Cancer Therapy; Cancer Treatment; Malignant Neoplasm Therapy; Malignant Neoplasm Treatment
Other: Health Care Delivery — Receive in home cancer treatment with CCBW
  Other Names: Care Delivery; Health Services Delivery, Other; Healthcare Delivery
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial evaluates the impact of cancer therapy in the patients' home compared to in the clinic on safety, side effects, patient preference, and satisfaction in Black men with prostate cancer that has spread to nearby tissue or lymph nodes (locally advanced), that has increasing prostate-specific antigen after treatment (biochemically recurrent) or that has spread from where it first started (primary site) to other places in the body (metastatic). Typically drug-related cancer care is conducted at a medical center which causes patients to have to spend considerable time away from family, friends, and familiar surroundings. This separation may add to the physical, emotional, social, and financial burden for patients and their families during this difficult time in their lives. Therapy administered to a patient in the patients' residence in the comfort of familiar surrounding using Cancer Connected Access and Remote Expertise (CARE) Beyond Walls (CCBW) may help reduce psychological and financial distress, increase access to care and improve treatment compliance. Giving cancer therapy in the home compared in the clinic may be safe, tolerable and improve patient satisfaction with overall cancer care in Black men with locally advanced, biochemically recurrent or metastatic prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish patient-centeredness by comparing patient ratings of their overall cancer care experience in the clinic versus in the home.

II. To establish patient-centeredness by evaluating patient preferences regarding the location of cancer treatment delivery.

SAFETY OBJECTIVES:

I. To assess the safety of home administered intravenous (IV)/subcutaneous (SQ) drug treatment by a home health provider with remote patient monitoring and Command Center support as measured by the incidence of grade 3+ adverse events at least possibly related to cancer treatment delivery.

II. To describe the incidence of acute care visits, emergency room visits, and hospitalizations during the entire study treatment period and by location of cancer treatment delivery (i.e., during in-clinic cancer treatment versus at-home cancer treatment).

III. To describe the incidence of avoidable (in the opinion of the treating physician) acute care visits, emergency room visits, and hospitalizations during at-home cancer treatment.

SECONDARY OBJECTIVE:

I. To evaluate the impact of home cancer treatment delivery on patient-reported function and global health/quality of life, patient-reported symptoms, satisfaction, and clinical outcomes.

EXPLORATORY OBJECTIVES:

I. To summarize patient perceptions and reasons for patient preferences regarding the location of cancer treatment delivery.

II. To describe overall survival. III. To assess the cost outcomes related to patient treatment in the clinic or in the home.

OUTLINE:

Patients receive standard of care treatment in the clinic for 6-12 weeks then receive treatment in the home with CCBW for 12-24 weeks in the absence of disease progression or unacceptable toxicity. Patients receive any remaining treatment in the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Participant must be receiving a standard-of-care treatment regimen listed in this protocol that is being used in accordance with standard medical practice. Specifically, it must be either a) FDA-approved for the participant's disease indication, or b) recommended in nationally recognized professional guidelines (e.g., NCCN, ASCO, ASH, etc.) as standard of care for the disease indication. Off-label use is permitted only if supported by such guidelines
* Black or African American male patients with locally advanced, high risk, biochemical recurrent, or metastatic prostate cancer who are currently receiving or planning to start treatment with one or more of the eligible regimens. Patients may be on any combination of these regimens, provided that at least one is administered by a home health nurse [co-administration with second generation antiandrogens, poly adenosine diphosphate-ribose polymerase (PARP) inhibitors, oral gonadotrophin releasing hormone (GnRh) antagonists, estrogens, or older antiandrogens are allowed but combinations of oral regimens only are not permitted]

  * Androgen deprivation therapy (ADT):

    * Leuprolide intramuscular (IM) or subcutaneous (SQ), 4 or 12 weeks cycle length
    * Degarelix SQ, 4 weeks cycle length
  * Chemotherapy: Cabazitaxel IV, 3 weeks cycle length
  * Immunotherapy: Pembrolizumab IV, 3 weeks cycle length
  * Bone modifying agent + any of the prostate cancer treatments:

    * Zoledronic acid IV, 4 or 12 weeks cycle length
    * Denosumab SQ, 4 or 12 weeks cycle length
* Patients who are anticipated to continue the treatment regimen they are currently prescribed for at least 18 weeks following registration (if on chemotherapy or immunotherapy) or 24 weeks following registration (for all other treatment regimens)
* Residing within the area serviced by supplier
* Provide written informed consent
* Willing and able to comply with the study protocol in the investigator's judgement
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1, or 2 for patients on any qualifying treatment (tx) regimen; ECOG PS 0, 1, 2, or 3 for patients on ADT with or without second generation antiandrogen
* Ability to complete questionnaire(s) by themselves or with assistance
* Willingness to follow birth control requirements for males of reproductive potential

Exclusion Criteria:

* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Current inpatient hospitalization (excluding admission to the Advanced Care at Home program)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Myocardial infarction ≤ 6 months
  * Wound healing disorder
  * Or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with any severe infection within 4 weeks prior to registration including, but not limited to, hospitalization for complications of infections should not be enrolled in the trial (in the current situation, this also applies to patients with suspected or confirmed COVID-19 infection)
* Anticipation of the need for major surgery during the course of study treatment

  * Note: Concomitant radiation therapy during the study period is allowed
* Not cleared for treatment in home via social stability screening
* Patients who received at home treatment through involvement in another CCBW trial

  * Note: Patients who enrolled in another CCBW trial but had to be withdrawn prior to initiating treatment in the home would still be eligible

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2028-08-27 (Estimated); Study Completion 2028-08-27 (Estimated)

PRIMARY OUTCOMES:
Patient rating of overall cancer care experience - CAHPS | Up to 48 weeks
  Patient rating of their overall cancer care experience after 12 weeks of at-home cancer treatment will be compared to the same rating after 6 or 12 weeks of in-clinic cancer treatment. Will be assessed using patient ratings from a single item from the Consumer Assessment of Healthcare Providers (CAHPS). Participants will rate "your overall cancer care experience" on a 0 to 10 scale where 0 is the worst experience possible and 10 is the best experience possible.
Patient preferences regarding the location of cancer treatment delivery | Up to 48 weeks
  Will be assessed by a single item asking patients to rate their preferred location for cancer treatment delivery on a 1 to 7 scale: 1=strongly prefer in clinic, 2=moderately prefer in clinic, 3=slightly prefer in clinic, 4=no preference, 5=slightly prefer at home, 6=moderately prefer at home, 7=strongly prefer at home.
Incidence of grade 3+ adverse events (AEs) | Up to 30 days after last dose of study treatment
  Incidence, type, and severity of AEs experienced during the study period will be reported. The maximum grade for each type of adverse event will be summarized using Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. For individual adverse events and overall, the frequency and proportion of grade 3+ adverse events and grade 3+ adverse events at least possibly related to cancer treatment delivery will be reported for the entire study treatment period and by location of cancer treatment delivery (i.e., in clinic versus at home).
Acute care visits, emergency room visits, and hospitalizations | Up to 48 weeks
  The frequency and proportion of patients who experience an acute care visit, emergency room visit, or hospitalization will be reported for the entire study treatment period and by location of cancer treatment delivery (i.e., during in clinic cancer treatment versus at-home cancer treatment).
Avoidable acute care visits, emergency room visits and hospitalizations | Up to 48 weeks
  The frequency and proportion of patients who experience an avoidable acute care visit, emergency room visit, or hospitalization while receiving at-home cancer treatment will be reported. Whether an acute care visit, emergency room visit, or hospitalization could have been avoided from changing the location of cancer treatment delivery will be in the opinion of the treating physician.

SECONDARY OUTCOMES:
Patient-reported function and global health status/quality of life | Up to 48 weeks
  Will be measured by the European Organization for the Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Functioning 17 (QLQ-F17), scored following its published scoring algorithm. Higher scores indicate better quality of life
Patient-reported symptoms as measured by Patient Reported Outcomes (PRO)-CTCAE | Up to 48 weeks
  PRO-CTCAE uses a 0-4 scoring system for most items, with 0 representing the absence of a symptom or no impact, and 4 representing the highest severity or impact. Some items, specifically those assessing presence, use a 0/1 (absent/present) scale. The frequency and proportion of patients with a maximum baseline-adjusted composite score ≥ 3 during the study treatment period and by location of cancer treatment delivery will be reported.
Patient-reported symptoms as measured by Functional Assessment of Cancer Therapy General Population 5 (FACT GP5) | Up to 48 weeks.
  The FACT GP5 consists of a single question, "I am bothered by side effects of treatment," rated on a scale of 0-4 where 0=not at all and 4=very much.
Patient Satisfaction and Feedback Questionnaire | Up to 48 weeks
  Patient satisfaction will be measured by the Patient Satisfaction and Feedback Questionnaire (specific to this study). The questionnaire consists of 30 questions evaluating different aspects of care, including level of care (excellent, very good, good, faire poor), preference for location of care (at home vs in clinic), comparison of care at home vs in clinic (strongly agree, disagree, neither agree nor disagree, agree, strongly agree), communication received from care team (0-10 where 0=worst communication possible and 10=best communication possible), transition to care at home and use of at-home equipment (very easy, easy, neither, difficult, very difficult). Patient responses will be summarized descriptively.
Patient satisfaction - Was It Worth It Questionnaire | Up to 48 weeks
  Will be measured by the Was It Worth It Questionnaire, which consists of 3 questions answered with yes/no/undecided, two questions answered on a e-point scale (better, same, worse), and one open-ended question (one things that could have been done to improve patient experience). Patient responses will be summarized descriptively.

CONTACTS AND LOCATIONS:
Overall Officials: Roxana S. Dronca, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials